CLINICAL TRIAL: NCT05015491
Title: A Single Arm Study to Assess the Effects of Online App Weight Loss Programs on Liver Health in Obese Adults
Brief Title: Effects of Online App Weight Loss Programs on Liver Health in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noom Inc. (Industry)
Collaborators: Arizona Liver Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Noom 2021-01
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: NASH; Fatty Liver; NAFLD; Weight Loss
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Noom Healthy Weight Program (Experimental): The Noom platform uses a cognitive behavioral approach to weight loss that integrates set content with interaction with live coaches to support client efforts at behavior change. The Healthy Weight program follows guidelines from the Obesity Society's "2013 Guidelines for the Management of Overweight and Obesity in Adults" NIH "Practical Guide on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults". It has 52 weeks of curriculum with 1-3 articles to read per day (Reading level: Grade 6-8).
  Interventions: Behavioral: Noom Healthy Weight Program

INTERVENTIONS:
Behavioral: Noom Healthy Weight Program — The Healthy Weight program follows guidelines from the Obesity Society's "2013 Guidelines for the Management of Overweight and Obesity in Adults" NIH "Practical Guide on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults". Users are encouraged to log their weight (Weight Logging) at least 1x/week and log their food and beverages (Food Logging) daily. Exercise logging (steps via automatic collection or manually added) is done daily. The Noom Food color grading system is founded on calorie-density (Volumetrics diet, Barbara Rolls) and is a simple and effective method for creating long lasting changes in diet and food choice. Coaches are contacted via In-app messaging or phone communication.

SUMMARY:
The primary objective of this trial is to assess the effects of online app weight loss programs on liver health in obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 years of age, inclusive, at Day -7.
* BMI of 30.00 to 49.99 kg/m2, inclusive, at Day -7.
* Has no plan to change smoking habits during the study period.
* Has ability to access study related online programs and apps.
* Willing to follow study instructions, as well as complete online questionnaires.
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigators, Sponsor and Collaborator.

Exclusion Criteria:

* Self-reported presence of uncontrolled cardiac, renal, endocrine, pulmonary, biliary, pancreatic, gastrointestinal, or neurological disorders or cancer (except for non-melanoma skin cancer) that may affect the subject's ability to adhere to the study protocol and/or affect study outcomes as assessed by the PI.
* Self-reported type 1 diabetes.
* History of gastrointestinal surgery for weight reducing purposes.
* Participation in a weight loss trial or a program/service intended to alter body weight (e.g., Noom, Weight Watchers); medications, dietary supplements or products that affect weight loss, nutrient absorption, appetite and satiety; or weight loss or gain ≥10 lb (4.5 kg) within 6 mo of Day -7.
* Extreme dietary habits (e.g., Atkins diet, very high protein, intermittent fasting) or eating disorder.
* Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded.
* Female with prior medical diagnosis of premenstrual syndrome or premenstrual dysphoric disorder.
* Unstable use of hormonal contraceptives, anti-hypertensive medication, medications for mental or emotional disorders, or thyroid hormones within 90 d of Day -7.
* Exposure to any non-registered drug product within 30 d of Day -7.
* Recent history of (within 12 mo of Day -7) or strong potential for alcohol or substance abuse. Alcohol abuse defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or

  1½ oz distilled spirits).
* ALT or AST > 5 x ULN at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Change in BMI | baseline to day 112
  BMI

SECONDARY OUTCOMES:
Fibroscan | Baseline to day 112
  Change in Controlled Attenuation Parameter (CAP) score CAP score is a measurement of fatty change in the liver. A CAP score is measured in decibels per meter (dB/m). It ranges from 100 to 400 dB/m.
Fibroscan - from baseline to day 112 | Baseline to day 112
  Change in Liver Stiffness Measurement (LSM)
Change Weight Efficacy Life-Style (WEL) subscale scores (negative emotion, availability, social pressure, physical discomfort, and positive activities) and a global score | Baseline to day 168
  This scale specifically evaluates self-efficacy judgments specific to eating behaviors in five situational factors: negative emotions, food availability, social pressure, physical discomfort, and positive activities. This measure has evidenced adequate psychometric properties, including internal consistency coefficients ranging from 0.76 to 0.90
Change in RAND-36 domain scores (emotional well-being, energy/fatigue, general health, pain, physical functioning, role limitations due to emotional problems, role limitations due to physical health, and social functioning). | Baseline to day 168
  The RAND 36-Item Health Survey (Version 1.0) laps eight concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. Scores represent the percentage of total possible score achieved.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Liver Health, Chandler, Arizona, United States

IPD SHARING:
Plan to Share IPD: No